CLINICAL TRIAL: NCT00815555
Title: CYP2D6 Genotyping by AmpliChipTM CYP450 for Tamoxifen-Treated Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 135/08
Record Dates: First submitted 2008-12-28; First posted 2008-12-30 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer
Keywords: receptor positive breast cancer; Tamoxifen treatment; CYP2D6 status; relapse
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women diagnosed with receptor positive breast cancer, treated with Tamoxifen
  Interventions: Other: There is no intervention - this is an observational study

INTERVENTIONS:
Other: There is no intervention - this is an observational study

SUMMARY:
The aim of the study is to examine whether tamoxifen-treated Israeli breast cancer patients who are CYP2D6 poor metabolizers (CYP2D6*4/*4 genotype) are at higher cancer relapse risk during 2.5-5-year follow-up period from initial diagnosis and primary treatment.

DETAILED DESCRIPTION:
Tamoxifen, the first-line drug for preventing breast cancer relapse, is typically prescribed for a 5-year follow-up period after diagnosis and primary treatment of estrogen receptor-positive breast cancer. Recent studies show that tamoxifen is only a pro-drug, while its major active metabolite, endoxifen, is formed in vitro by the liver enzyme CYP2D6. Preliminary observations from the US and Italy have suggested that tamoxifen is less efficacious for cancer relapse prevention in patients with deficient CYP2D6 activities. The FDA is currently reviewing the new data and is likely to modify the tamoxifen label accordingly. It was suggested that an aromatase inhibitor drug such as letrozole might be more beneficial for these patients.

The proposed study would retrospectively test CYP2D6 genotypes in 200 - 300 estrogen receptor (ER) positive breast cancer patients who are treated with tamoxifen post-operatively. Blood collected with informed consent would be used for examining the patients CYP2D6 genotype, and identifying those who are CYP2D6 poor metabolizers (CYP2D6*4/*4 genotype), and for measurement of endoxifen blood level in those women who are on the drug.

AmpliChipTM CYP450 is a microarray chip which contains millions of tiny DNA molecules, providing comprehensive coverage of gene variations that play a role in the metabolism of approximately 25% of all prescription drugs. The AmpliChipTM CYP450 test is intended to be an aid for physicians in individualizing treatment doses for patients receiving therapeutics metabolized through these enzymes.

The clinical data collected would examine if these individuals, as well as those treated with CYP2D6 inhibiting drugs such as paroxetine and fluoxetine, have higher cancer relapse rates.

The study, combined with similar findings from other countries, and possibly integrated later on with an international network study, would be imperative for modifying treatment recommendations for breast cancer therapy. Specifically, if the US and Italian findings are confirmed, it might be advisable to switch the 5-year follow-up treatment for breast cancer patients with ER positive primary tumors who are CYP2D6 poor metabolizers from tamoxifen to an aromatase inhibitor drug such as letrozole.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18
* Treated with Tamoxifen following diagnosis of breast cancer

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with receptor positive breast cancer, treated with Tamoxifen
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Tamoxifen efficacy for avoiding breast cancer relapse in relation to CYP2D6 genotype

SECONDARY OUTCOMES:
Prevalence of CYP2D6 poor metabolizers genotype in Israeli female population treated with Tamoxifen

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Unit - Assaf Harofeh Medical Center, Ẕerifin, Israel